CLINICAL TRIAL: NCT01386125
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of 200 mcg BID Mometasone Furoate Nasal Spray (MFNS) in the Treatment of Nasal Polyps (Protocol No. P05604)
Brief Title: A Study of the Effectiveness and Safety of Mometasone Furoate Nasal Spray (MFNS, SCH 032088) for the Treatment of Nasal Polyps (P05604)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05604
Record Dates: First submitted 2011-06-09; First posted 2011-06-30 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2022-02

CONDITIONS: Nasal Polyps
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mometasone Furoate Nasal Spray (MFNS) (Experimental): Participants receive mometasone furoate nasal spray (MFNS) 200 mcg twice daily (BID) for 16 weeks
  Interventions: Drug: Mometasone Furoate Nasal Spray (MFNS)
- Placebo (Placebo Comparator): Participants receive matching placebo nasal spray BID for 16 weeks
  Interventions: Drug: Placebo for MFNS

INTERVENTIONS:
Drug: Mometasone Furoate Nasal Spray (MFNS) — MFNS, 200 mcg BID administered as two 50 mcg sprays in each nostril BID for up to 16 weeks
  Arms: Mometasone Furoate Nasal Spray (MFNS)
Drug: Placebo for MFNS — Two sprays in each nostril BID for up to 16 weeks
  Arms: Placebo

SUMMARY:
This study will evaluate the effectiveness and safety of MFNS in improving nasal congestion/obstruction and in reducing bilateral nasal polyps.

ELIGIBILITY:
Inclusion Criteria:

* Must be Chinese
* Must have a diagnosis of bilateral nasal polyps
* Clinically significant nasal congestion/obstruction must be present
* Must be in good health, free of any clinically significant disease that would interfere with the study schedule or procedures, or compromise the participant's safety
* Must have negative urine pregnancy test
* Must be using or agree to use a medically accepted method of contraception prior to Screening and during the study

Exclusion Criteria:

* Have a history of seasonal allergic rhinitis within the last two years
* Have had sinus or nasal surgery within the past six months
* Have presumed fibrotic nasal polyps
* Have had three or more nasal surgeries
* Have had any surgical procedure that prevents an accurate grading of the polyps
* Complete (or near complete) nasal obstruction
* Have acute sinusitis, concurrent nasal infection or have had a nasal infection within two weeks
* Have ongoing rhinitis medicamentosa
* Have Churg Strauss syndrome (vasculitis, asthma, fever, and eosinophilia)
* Have dyskinetic ciliary syndromes, eg, Young's syndrome (sinopulmonary infections and obstructive azoospermia) or Kartagener's syndrome (immobile cilia)
* Have been treated within the last 4 weeks with intranasal steroids
* Have used any investigational drug in the last 30 days
* Have a hypersensitivity to corticosteroids or are allergic to aspirin
* Have an ongoing upper respiratory tract infection or had an upper respiratory tract infection within two weeks
* Have a nasal septal deviation needing corrective surgery
* Have a nasal septal perforation
* Have asthma that required in-patient hospitalization for asthma control within six months, required ventilator support for respiratory failure secondary to their asthma within the last five years, required admission to the hospital for management of airway obstruction on two or more occasions within the past year, or required use of more than 14 days of systemic steroid use in previous six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 748 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhou B, He G, Liang J, Cheng L, Mehta A, Liu S, Yu W, Wang Z, Han D. Mometasone furoate nasal spray in the treatment of nasal polyposis in Chinese patients: a double-blind, randomized, placebo-controlled trial. Int Forum Allergy Rhinol. 2016 Jan;6(1):88-94. doi: 10.1002/alr.21650. Epub 2015 Nov 17. PMID 26575524

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Started | 375 | 373
Completed | 350 | 336
Not Completed | 25 | 37
Not completed — Lost to Follow-up | 3 | 9
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 5 | 7
Not completed — Disease Progress | 1 | 2
Not completed — Withdrawal by Subject | 13 | 12
Not completed — Adverse Event | 2 | 5
Not completed — Lack of Efficacy | 0 | 1
Not completed — Participant Leaving Country | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- MFNS: Participants receive MFNS 200 mcg BID for 16 weeks
- Total: Total of all reporting groups
Arm/Group | MFNS | Placebo | Total
Number analyzed (Participants) | 375 | 373 | 748
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (13.49) | 46.8 (13.75) | 46.8 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 134 | 285
  Male | 224 | 239 | 463

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Congestion/Obstruction Score
Description: At Baseline, the Investigator and participant jointly evaluated the signs and symptoms of congestion/obstruction. After Baseline, participants scored the signs and symptoms of congestion/obstruction every morning immediately prior to dosing using a morning instantaneous congestion/obstruction score. This score reflected the participant's condition at that time (instantaneous) and ranged from 0 to 3 (0=none, 1=mild, 2=moderate, 3= severe), with a lower score indicating less congestion/obstruction. Congestion/obstruction scores were averaged over Weeks 1-4 of the treatment period. Data are compared using Least Square (LS) Means. LS Mean Change from Baseline = LS Mean Score averaged over Weeks 1-4 - LS Mean Score for Baseline.
Time Frame: Baseline and Weeks 1-4
Population: The Full Analysis Set (FAS) population consisted of all randomized participants who received at least one dose of study treatment and who had a baseline and at least one post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MFNS | Placebo
Number analyzed (Participants) | 372 | 371
score on a scale | -0.56 (0.03) | -0.42 (0.03)
Statistical Analysis 1: Comparison: MFNS vs Placebo; Test type: Superiority or Other; p = 0.0007, ANCOVA; Difference in LS Means = -0.14, 95% CI 2-sided [-0.22 to -0.06]

2. Primary Outcome: Change From Baseline in Total Polyp Size Score
Description: An endoscopic nasal examination was performed by the Investigator. Bilateral nasal polyps were scored as follows for each notril (left and right): 0=no polyps, 1=polyps in middle meatus not reaching below inferior border of middle turbinate, 2=polyps reaching below inferior border of middle turbinate but not inferior border of inferior turbinate, 3=large polyps reaching to or below the lower borders of the inferior turbinate or polyps medial to the middle turbinate. Total polyp size score ranged from 0 to 6 (scored 0 to 3 for each nostril), with a lower score indicating smaller-sized polyps. LS Mean Change from Baseline = LS Mean Score for Week 16 - LS Mean Score for Baseline.
Time Frame: Baseline and Week 16
Population: The FAS population consisted of all randomized participants who received at least one dose of study treatment and who had a baseline and at least one post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MFNS | Placebo
Number analyzed (Participants) | 375 | 373
score on a scale | -0.76 (0.05) | -0.45 (0.05)
Statistical Analysis 1: Comparison: MFNS vs Placebo; Test type: Superiority or Other; p < 0.0001, Constrained longitudinal data analysis; Difference is LS Means = -0.30, 95% CI 2-sided [-0.45 to -0.15]

ADVERSE EVENTS:
Time Frame: Up to approximately 20 weeks
Arm/Group | MFNS | Placebo
Serious Adverse Events (participants affected / at risk) | 2/375 | 3/373
Other Adverse Events (participants affected / at risk) | 0/375 | 0/373
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MFNS (N=375) | Placebo (N=373)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.